CLINICAL TRIAL: NCT07165665
Title: The Effect of Nervus Vagus Stimulation on Spasticity, Autonomic Function, Motor Function and Quality of Life in Children With Spastic Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Server ERDOĞMUŞ, Msc. PT. / Research Assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-60116787-020-729758
Record Dates: First submitted 2025-08-26; First posted 2025-09-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Children With Cerebral Palsy
Keywords: Cerebral palsy; Children; Nervus vagus; autonomic nervous system; Quality of life; Motor function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: In this study, the effects on spasticity, autonomic function, motor function, and quality of life in children with spastic cerebral palsy will be examined. The children will be divided into two groups:
  Bobath Group: Only the Bobath (Neurodevelopmental Treatment) approach will be applied.
  Bobath+ VNS Group: Non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) will be applied in addition to the Bobath approach.
  Both groups will receive treatment twice a week for 8 weeks, and spasticity, motor function, autonomic function, and quality of life will be assessed before and after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath+ VNS Group (Experimental): Non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) will be applied in addition to the Bobath approach.
  Interventions: Other: Bobath (Neurodevelopmental Treatment) approach; Device: Non-invasive transcutaneous auricular vagus nerve stimulation (taVNS)
- Bobath Group (Experimental): Only the Bobath (Neurodevelopmental Treatment) approach will be applied.
  Interventions: Other: Bobath (Neurodevelopmental Treatment) approach

INTERVENTIONS:
Other: Bobath (Neurodevelopmental Treatment) approach — The control group will receive only the standard Bobath (Neurodevelopmental Treatment, NDT) approach.
Device: Non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) — The intervention group will receive the standard Bobath (Neurodevelopmental Treatment, NDT) approach combined with non-invasive transcutaneous auricular vagus nerve stimulation (taVNS).
  Arms: Bobath+ VNS Group

SUMMARY:
Introduction:

Cerebral palsy (CP) is a heterogeneous neurodevelopmental syndrome affecting muscle tone, motor skills, and movement due to brain injury during developmental stages. The etiology of CP is associated with factors such as prematurity, low birth weight, and pregnancy or birth complications. The spastic type is the most common motor disorder, characterized by increased reflexes and muscle hypertonia in the extremities. Spasticity arises from upper motor neuron lesions, leading to dysregulation in spinal and brain pathways (corticospinal, reticulospinal, vestibulospinal) and involves complex modulation of muscle tone and stretch reflexes.

The autonomic nervous system regulates visceral functions, while the vagus nerve, through its parasympathetic fibers, exerts widespread influence on the heart, respiratory system, and gastrointestinal system. It controls organ function via motor, sensory, and parasympathetic fibers originating from three medullary nuclei (nucleus ambiguus, dorsal motor nucleus, and nucleus solitarius). Vagus nerve stimulation (VNS) modulates the central nervous system by stimulating afferent fibers, increasing GABA and other inhibitory neurotransmitter levels, reducing excitatory signals, and potentially influencing spasticity. VNS can be applied invasively or non-invasively (transcutaneous VNS, tVNS); particularly, tVNS applied to the left ear is a safe and well-tolerated method with therapeutic potential in epilepsy and motor disorders.

This study aims to investigate the effects of non-invasive auricular vagus nerve stimulation (taVNS) combined with the Bobath approach on motor function, autonomic function, spasticity, activities of daily living, and quality of life in children with spastic cerebral palsy (CP).

Materials and Methods:

Planned as a prospective, controlled study, children with CP will be randomly assigned to two groups. The intervention group will receive the standard Bobath program administered by physiotherapists with at least 3 years of experience, combined with transcutaneous auricular vagus nerve stimulation (taVNS). The control group will receive only the Bobath approach. Both groups will undergo therapy twice a week for 8 weeks.

Outcome Measures:

Motor function: Assessed using the Gross Motor Function Measure (GMFM-88) and the Gross Motor Function Classification System (GMFCS).

Spasticity: Measured with the Modified Ashworth Scale (MAS).

Quality of life: Evaluated using the Pediatric Quality of Life Inventory (PedsQL).

Autonomic function: Heart rate variability (HRV) analyzed using the Elite HRV Corsense device. Measured parameters include RMSSD, LF power, HF power, LF/HF ratio, and mean heart rate.

Inclusion Criteria:

Diagnosis of spastic cerebral palsy

Aged 8-18 years

MAS score between 1 and 3

GMFCS Level I-III

Adequate cognitive level

No previous vagus nerve stimulation

No cardiovascular or chronic respiratory disease

Informed consent from parent/legal guardian

Exclusion Criteria:

Severe cardiovascular or pulmonary disease

Respiratory failure requiring mechanical ventilation

History of epilepsy or active seizures

MAS 0 or 4, GMFCS IV-V

Skin conditions in the neck/ear region preventing stimulation

Inability to obtain sufficient consent or perform assessments

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic cerebral palsy
* Aged between 8 and 18 years
* No chronic respiratory or cardiovascular disease
* Having spasticity between 1 and 3 according to the Modified Ashworth Scale (MAS)
* Classified as Level I-III according to the Gross Motor Function Classification System (GMFCS)
* Sufficient cognitive ability to participate in the study and complete assessments
* No previous vagus nerve stimulation and no contraindications for the procedure
* No congenital or acquired cardiovascular disease
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* History of congenital or acquired severe cardiovascular or pulmonary disease
* Requirement of mechanical ventilation due to respiratory failure
* History of epilepsy or active seizures
* Previous vagus nerve stimulation
* Inability to complete assessments due to severe cognitive impairment
* Having spasticity of 0 or 4 according to the Modified Ashworth Scale (MAS)
* Classified as Level IV-V according to the Gross Motor Function Classification System (GMFCS)
* Presence of skin disease in the neck or ear region or any condition preventing vagus nerve stimulation
* Inability to obtain parental/legal guardian consent for participation in the study

Withdrawal Criteria for Participants:

Participants will be withdrawn from the study if they are unable to complete the administered tests, assessments, or questionnaires.

Study Termination Criteria:

The study will be concluded once the planned sample size has been reached.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Demographic Data | A pre-test will be conducted to determine participants' baseline levels before the intervention; assessments will be repeated at 8 weeks (post-intervention) to evaluate changes.
  Demographic Data Form: Sociodemographic data form will be created for the patients.
Motor Function | A pre-test will be conducted to determine participants' baseline levels before the intervention; assessments will be repeated at 8 weeks (post-intervention) to evaluate changes.
  GMFM-88: A scale consisting of 88 items across 5 subscales, used to assess gross motor functions in children. Scoring is done using a 0-3 Likert scale, and the average of the percentage scores for each subscale is calculated to obtain the total score.
Motor Function Classification | A pre-test will be conducted to determine participants' baseline levels before the intervention; assessments will be repeated at 8 weeks (post-intervention) to evaluate changes.
  GMFCS: Classifies the motor function levels of children with CP into 5 levels.
Spasticity | A pre-test will be conducted to determine participants' baseline levels before the intervention; assessments will be repeated at 8 weeks (post-intervention) to evaluate changes.
  MAS: Assesses the degree of spasticity on a scale from 0 to 4.
Children's Quality of Life | A pre-test will be conducted to determine participants' baseline levels before the intervention; assessments will be repeated at 8 weeks (post-intervention) to evaluate changes.
  PedsQL (Children's Quality of Life Scale): Measures quality of life in children aged 2-18, covering physical, emotional, social, and school functioning. Scores are linearly converted to a 0-100 scale.
Autonomic Function | A pre-test will be conducted to determine participants' baseline levels before the intervention; assessments will be repeated at 8 weeks (post-intervention) to evaluate changes.
  Autonomic Function: Parasympathetic and sympathetic activities will be measured using HRV analyses

CONTACTS AND LOCATIONS:
Overall Officials: ERDOĞAN KAVLAK, PROF. DR., Study Director
Locations (1):
- VM Medical Park Bursa Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No